CLINICAL TRIAL: NCT03926000
Title: The Effect of Pregabalin Premedication on Anaesthetic Requirements and Recovery Time After Knee Arthroscopy
Brief Title: Pregabalin Premedication for Knee Arthroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Dr Ezzeldin Ibrahim, Professor, Menoufia University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: MenoufiaU2019/7
Record Dates: First submitted 2019-04-22; First posted 2019-04-24 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Knee Arthroscopy
MeSH Terms: interventions — Pregabalin; Premedication

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregabalin (PG) (Active Comparator): Patients will receive 150 mg pregabalin one hour before the procedure.
  Interventions: Drug: Pregabalin (PG)
- Control placebo (C) (Placebo Comparator): Patients will receive placebo tablet one hour before surgery.
  Interventions: Drug: Control placebo (C)

INTERVENTIONS:
Drug: Pregabalin (PG) — Pregabalin 150 mg one hour before the procedure as premedication.
  Other Names: Pregabalin for premedication
  Arms: Pregabalin (PG)
Drug: Control placebo (C) — Placebo tablets one hour before the procedure as premedication.
  Other Names: Placebo for premeditation.
  Arms: Control placebo (C)

SUMMARY:
Outpatient arthroscopic knee surgery can be performed with general or regional anesthesia. Recent data suggest that spinal and epidural anesthesia require longer discharge times than the newer shorter-acting general anesthetic drugs. Ideal premedication drug should relieve anxiety, produce amnesia and sedation, decrease secretions, prevent nausea and vomiting, have dose sparing effect on the anaesthetic drugs, and suppress pressor response to laryngoscopy and intubation. Recently, gabapentin and pregabalin were suggested as pre-operative drugs to decrease anxiety, stress response to laryngoscopy and post operative pain.

DETAILED DESCRIPTION:
112 patients undergoing elective knee arthroscopy will randomly divided into two equal groups, 56 patients each. All patients will receive premedication one hour before the procedure. PG group will receive 150 mg pregabalin and C group will receive placebo. All patients will receive total intravenous anesthesia to achieve optimum working conditions. Intra-operative total amount of anesthetics will be compared in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective knee arthroscopy.
* Patients aged between 21 and 50 years old.
* Patients with American Society of Anaesthesiologists physical status I or II.

Exclusion Criteria:

* Patients with known allergy to any drug used in the study.
* Patients with chronic use of analgesics and/or sedatives.
* Patients with sleep apnea syndrome.
* Patients with renal or hepatic dysfunction.
* Patients with psychiatric disorders.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Total amount of anesthetics | 45 minutes during the procedure
  Total amount of anesthetics used during the procedure.

SECONDARY OUTCOMES:
Patients' satisfaction: satisfaction score | 30 minutes after the end of the procedure
  Patient's satisfaction score will be recorded using a score ranging from 0 not satisfied and 5 totally satisfied. The score will be done using a questioner designed by the researchers.